CLINICAL TRIAL: NCT04739852
Title: The Kinetics of Autophagy During Periodic Fasting in Healthy People and Patients With Rheumatoid Arthritis or Metabolic Syndrome - an Exploratory Clinical Study
Brief Title: An Exploratory Clinical Study on Autophagy During Fasting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Klinik und Poliklinik für Psychiatrie und Psychotherapie, Universitätsklinikum Bonn AöR (Unknown)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Autophagy Fasting
Record Dates: First submitted 2021-01-05; First posted 2021-02-05 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Arthritis, Rheumatoid; Syndrome, Metabolic; Healthy
Keywords: Fasting; Autophagy
MeSH Terms: conditions — Arthritis, Rheumatoid; Metabolic Syndrome; Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: 3 groups of different inclusion criteria (healthy, metabolic syndrome or rheumatoid arthritis) undergoing the same intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Participants (Active Comparator): Healthy participants
  Interventions: Other: Fasting
- Metabolic Syndrome (Active Comparator): Participants with diagnosed metabolic syndrome
  Interventions: Other: Fasting
- Rheumatoid Arthritis (Active Comparator): Participants with diagnosed rheumatoid arthritis
  Interventions: Other: Fasting

INTERVENTIONS:
Other: Fasting — Patients undergo a 5-10 day fasting period with a dietary energy supply 350-400kcal per day with fruit and vegetable juices or, if not feasible, an established fasting-mimicking diet of 600-800 kcal according to Longo et al.

SUMMARY:
Autophagy is considered one of the key molecular mechanisms for the broad preventive and therapeutic effects of periodic fasting. While it is generally known that fasting induces autophagy, there are no human studies that focus on the size and temporal kinetics of autophagy and its association with fasting specific signaling pathways. The kinetics of autophagy in patients with chronic diseases will now be compared with the kinetics of autophagy in healthy subjects, who both fast according to the same scheme; and further changes in metabolic and inflammatory parameters will be investigated.

DETAILED DESCRIPTION:
Therapeutic fasting has been used for many decades in naturopathy and integrative medicine clinically successfully in the treatment of chronic diseases and pain syndromes. In particular, fasting therapy is used for chronic rheumatic, inflammatory, and metabolic diseases with increasing patient demand in specialized clinical facilities (fasting clinics).

Within the various historically developed forms of fasting, the fasting program according to the Buchinger Wilhelmi method has established itself worldwide as the most frequently applied method. This involves a subtotal caloric restriction with a daily caloric intake (200-400kcal/day) in the form of liquid components over a defined period of at least 10 days, accompanied by supporting measures of a health-promoting lifestyle program with elements such as exercise therapy, manual procedures, stress reduction and hydro-balneotherapy.

In early randomized studies and a systematic review, the effectiveness of inpatient fasting therapy for patients with rheumatoid arthritis was proven with 1a evidence. For the other indications, there is mainly empirical evidence or data from observation or prospective uncontrolled studies. In recent years, extensive basic science research activity has developed in the area of caloric restriction and intermittent fasting. In this context, a large number of favorable animal experimental findings have been demonstrated by defined fasting periods, including reductions in insulin, IGF-1, increases in adiponectins, insulin sensitivity, neurotrophic factors, and, over longer observation periods, a decrease in the incidence of cardiovascular, inflammatory, and metabolic, and more recently oncological diseases in a wide variety of animal species.

Numerous experimental studies have demonstrated that fasting or total or subtotal caloric restriction is a potent inducer of cellular autophagy. For autophagy, numerous beneficial effects on chronic diseases or disease defense functions have now been experimentally documented and also hypothesized for humans, including neurodegenerative and metabolic diseases, but also acute infections and inflammatory diseases. Unclear to date is the kinetics of the autophagy enhancing effect of fasting. In theoretical transfer from animal experimental data, an increase is postulated between 12 and 36h of fasting and possibly a decrease after several days.

Against this background, autophagy will now be investigated for the first time in blood samples from fasting healthy and diseased individuals in an exploratory clinical study.

ELIGIBILITY:
Inclusion Criteria:

* One of the following diagnoses: rheumatoid arthritis, metabolic syndrome OR healthy volunteer
* Beginning (first 24h) inpatient treatment or hospital stay at Immanuel Hospital Berlin, Department of Naturopathy OR healthy volunteer
* Present written declaration of consent

Exclusion Criteria:

* Insufficient linguistic communication
* Dementia or other cognitive disorder
* Pregnancy or lactation
* Simultaneous participation in another clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Exploratory Proteomics of Autophagy Processes I | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  - Change in protein levels of autophagy biomarkers (LC3II & p62) of isolated PBMCs (peripheral blood mononuclear cells) by Western Blotting, change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
Exploratory Proteomics of Autophagy Processes II | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  - Change in protein levels and protein phosphorylation by untargeted mass spectrometry-based proteomics and phosphoproteomics of isolated PBMCs (peripheral blood mononuclear cells), change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up

SECONDARY OUTCOMES:
Muscle mass | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Estimation of the body composition via bio-electrical impedance analysis (muscle mass in kg)
Body fat | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Estimation of the body composition via bio-electrical impedance analysis (body fat and visceral fat in %)
Resting blood pressure | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
Cutaneous carotenoid level (CCL) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Cutaneous carotenoid level (CCL), correlating with the overall antioxidant status, measured with a noninvasive skin carotenoid sensor (Biozoom®)
Heart rate | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
Waist to Hip Ratio | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
Body Mass Index (kg/m2) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
Disease Activity Score 28 (DAS-28-CRP) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Change from Baseline in the DAS-28-CRP, range from 2.0 to 10.0 while higher values meaning a higher disease activity and below of 2.6 meaning remission
Health Assessement Questionnaire (HAQ) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Change from Baseline in the HAQ, range from 0 to 3 while higher values meaning a higher grade of disability
Simplified Disease Activity Index Score (SDAI) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Change from Baseline in the SDAI, range from 0 to 86 with assumed range from 0.1 to 10mg/dL for CRP. Higher values mean a higher disease activity and below of 34 meaning remission.
Stress questionnaire (Cohen Perceived Stress Scale, CPSS) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Change from Baseline in the CPSS, range from 0 to 4 in each item. Scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the positively stated items and then summing across all scale items, higher values meaning a higher grade of perceived stress.
Mindful Attention Awareness Scale (MAAS) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Assessing full scale, range from 15 to 90, higher score values meaning a better outcome.
Numerical Analog Scales | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Assessing stress, back pain, headache, shoulder/neck tension, sleep quality and duration, exhaustion, nervousness, digestive complaints, mood on 0-10 points each.
Quality of Life questionnaire (WHO-5) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Change from Baseline in the WHO-5, range from 0 to 100 %, higher values meaning a higher grade of well-being
Hospital Anxiety and Depression Scale (HADS) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Assessing full scale, range 0-42, lower score meaning a better outcome
General Self-efficacy Short Scale (ASKU) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Assessing full scale, range 3-15, higher score meaning a better outcome
Mood questionnaire (Profile of Mood States, POMS) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Change from Baseline in Emotional Distress will be measured using the German Version of the Profile of Mood States (ASTS) short version (19 items, 7-point Likert scale; 0=not at all, 6=extremely). Lower scores indicate more stable mood profiles.
Sociodemographic Measurements | Day 1 (baseline)
  Age, gender, education level, household income, employment status, marital status, language spoken, complete family history, current and previous illness and co-morbidities, and current medications
Behavioral Factors | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Physical inactivity, coffee, health promoting activities via Likert Scales, range from 0 to 5 while higher values meaning a higher grade of agreement
Behavioral Factors: alcohol consumption | Day 1 (baseline), after 2 and 6 weeks
  Number of alcoholic beverages on average per week in the last month
Behavioral Factors: smoking | Day 1 (baseline), after 2 and 6 weeks
  Number of cigarettes on average per week in the last month
Behavioral Factors: fasting experience | Day 1 (baseline)
  Type, definition, duration and date of previous fasting experiences
Expectation questions | Day 1 (baseline)
  For fasting on a 5-point likert scale from 1 (nothing at all) to 5 (very strong)
Creatinine in µmol per liter (µmol/L) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
Estimated glomerular filtration rate (eGFR) in milliliter per minute (mL/min) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
Electrolytes | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  potassium (mmol/L) sodium (mmol/L)
Blood lipids and fasting glucose | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  triglycerides (mmol/L) total cholesterol (mmol/L) LDL (mmol/L) HDL (mmol/L) fasting glucose (mmol/L)
Insulin (mU/L) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
ß-Hydroxybutyrate | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Evaluate change in ketone body production by POCT
CrP (mg/L) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Evaluate change in CrP levels in participants with RA
Erythrocyte sedimentation rate (ESR) in millimeters per hour (mm/h) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Evaluate change in ESR in participants with RA
Rheumatoid factor (RF, IgM) (U/mL) | Day 1 (baseline)
  Evaluate RF status in participants with RA
Anti-cyclic citrullinated peptide (ACPA) (U/mL) | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Evaluate change in ACPA levels in participants with RA
Metabolic processes | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Targeted and quantitative analysis by mass spectrometry of change in metabolites of plasma, change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
Lipid profiling | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Targeted and quantitative analysis by mass spectrometry of change in plasma lipids, change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
Transcription expression patterns | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Change of the gene expression profile by RNA sequencing of isolated PBMCs (peripheral blood mononuclear cells), change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
Proteome/phosphoproteome/ubiquitinome patterns | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Evaluate proteome expression patterns through blood based proteome, phosphoproteome, and ubiquitinome analysis assessed prior to intervention (pre) vs. after 5-day fasting, day 2 of refeeding and 7 days post intervention
Epigentic patterns | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Evaluate epigentic methylation patterns through blood based epigenome analysis assessed prior to intervention (pre) vs. after 5-day fasting, day 2 of refeeding and 7 days post intervention
Exosomal protein patterns | change from baseline over 5 fasting days, to day 3 refeeding and to 7 days follow up
  Evaluate exosomal protein content through blood based metabolome analysis assessed prior to intervention (pre) vs. after 5-day fasting, day 2 of refeeding and 7 days post intervention

OTHER OUTCOMES:
Final questionnaire to record tolerability of fasting and nutrition, adverse effects | After 6 weeks
  Measurement of tolerability of fasting and nutrition as well as adverse effects via Likert Scales, range from 0 to 5 while higher values meaning a higher grade of agreement

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charite - Universitätsmedizin Berlin; Nils Gassen, Dr., Study Director — Department of Psychiatry and Psychotherapy University Bonn, Clinical Centre
Locations (1):
- Hochschulambulanz für Naturheilkunde der Charité-Universitätsmedizin Berlin am Immanuel-Krankenhaus, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No